CLINICAL TRIAL: NCT01125033
Title: Efficacy of Vitamin C, Vitamin E and Their Combination for Treatment of Restless Legs Syndrome in Hemodialysis Patients: a Randomized Double-blind, Placebo-controlled Trial
Brief Title: Study of Vitamin C, Vitamin E and Their Combination to Treat Restless Legs Syndrome in Hemodialysis Patients
Acronym: ShirazUMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Vice Chancellor for Research At Shiraz University of Medical Sciences, Shiraz Nephro-Urology Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 86-3893
Record Dates: First submitted 2010-05-14; First posted 2010-05-18 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Restless Legs Syndrome; Kidney Failure, Chronic
Keywords: Dialysis, Restless legs syndrome, Ascorbic acid, Vitamin E
MeSH Terms: conditions — Restless Legs Syndrome; Kidney Failure, Chronic | interventions — Ascorbic Acid; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin C & Vitamin E. (Experimental): The patients in this arm received one tablet of vitamin C (200 mg) and one capsule of vitamin E (400 mg) daily for 8 weeks
  Interventions: Drug: Vitamin C & Vitamin E
- Vitamin C & Placebo (Experimental): The patients in this arm received one tablet of vitamin C (200 mg) and one placebo capsule daily for 8 weeks.
  Interventions: Drug: Vitamin C
- Vitamin E & Placebo (Experimental): The patients in this arm received one capsule of vitamin E (400 mg) and one placebo tablet daily for 8 weeks.
  Interventions: Drug: Vitamin E
- Double Placebo (Placebo Comparator): The patients in this arm received one placebo capsule and one placebo tablet daily for 8 weeks.
  Interventions: Drug: Vitamin C Placebo & Vitamin E Placebo

INTERVENTIONS:
Drug: Vitamin C & Vitamin E — The patients in this arm received one tablet of vitamin C (200 mg) and one capsule of vitamin E (400 mg) daily for 8 weeks
  Arms: Vitamin C & Vitamin E.
Drug: Vitamin C — The patients in this arm received one tablet of vitamin C (200 mg) and one placebo capsule daily for 8 weeks.
  Arms: Vitamin C & Placebo
Drug: Vitamin E — The patients in this arm received one capsule of vitamin E (400 mg) and one placebo tablet daily for 8 weeks.
  Arms: Vitamin E & Placebo
Drug: Vitamin C Placebo & Vitamin E Placebo — The patients in this arm received one placebo capsule and one placebo tablet daily for 8 weeks.
  Arms: Double Placebo

SUMMARY:
The purpose of this study is to determine whether vitamin C, vitamin E and their combination are effective in the treatment of RLS in hemodialysis patients.

DETAILED DESCRIPTION:
RLS is a common problem in hemodialysis patients; 20 to 40% of hemodialysis patients suffer from RLS. Hemodialysis patients have a high oxidative stress status. Oxidative stress has been proposed to play an important role in the pathogenesis of RLS. Vitamin C and vitamin E are potent antioxidant agents that have already been shown to be effective in the treatment of periodic limb movement disorder (PLMD) in hemodialysis patients. PLMD is closely associated with RLS in hemodialysis patients. The aim of this study was to evaluate the efficacy of vitamin C, vitamin E and their combination in the treatment of RLS in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill Restless leg syndrome international criteria(IRLSSG)
* Patients who are stable on HD without any internment illness or admission

Exclusion Criteria:

* Patients who have renal stone
* Patients who receive medications with RLS aggravating or alleviating properties

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Absolute Change in IRLS Sum Score | 8 Weeks
  Absolute Change in IRLS Sum Score from Baseline to the End of Treatment Phase in Intention-to-treat Population

SECONDARY OUTCOMES:
Number of participants with adverse events | 8 Weeks
  Number of participants with adverse events throughout the treatment phase of the study would be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hamideh Akbari, MD, Principal Investigator — Shiraz University of Medical Sciences; Mohammad Mahdi Sagheb, MD, Study Chair — Shiraz University of Medical Sciences; Sahar Sohrabi Nazari, MD, Principal Investigator — Shiraz University of Medical Sciences; Mohammad Kazem Fallahzadeh, MD, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745